CLINICAL TRIAL: NCT02437253
Title: Pilot Study of the Effect of Adalimumab on Physical Function and Musculoskeletal Disease in Mucopolysaccharidosis Types I, II and VI
Brief Title: Effects of Adalimumab in Mucopolysaccharidosis Types I, II and VI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30535
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-05

CONDITIONS: Mucopolysaccharidosis Type I; Mucopolysaccharidosis Type II; Mucopolysaccharidosis Type VI
Keywords: Mucopolysaccharidosis; Inflammation; Tumor necrosis factor - alpha inhibitor
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI; Mucopolysaccharidoses; Inflammation | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab first, then Placebo (Experimental): Participants first received Adalimumab 20 mg subQ every other week (weight 15 to <30 kg) or 40 mg subQ every other week (weight ≥30 kg) for 16 weeks. Participants then received Placebo saline subQ (volume matching Adalimumab 20 mg or 40 mg subQ) every other week for 16 weeks.
  Interventions: Drug: Adalimumab; Other: Placebo
- Placebo first, then Adalimumab (Experimental): Participants first received Placebo saline subQ (volume matching Adalimumab 20 mg or 40 mg subQ) every other week for 16 weeks. Participants then received Adalimumab 20 mg subQ every other week (weight 15 to <30 kg) or 40 mg subQ every other week (weight ≥30 kg) for 16 weeks.
  Interventions: Drug: Adalimumab; Other: Placebo

INTERVENTIONS:
Drug: Adalimumab — Subjects will be treated with adalimumab (20 mg [weight 15-<30 kg] or 40 mg [weight ≥30 kg] administered subcutaneously [subQ] every other week) or placebo for 16 weeks, then cross-over to the other group for 16 weeks.
  Other Names: Humira
Other: Placebo — Saline placebo

SUMMARY:
The purpose of the study is to collect preliminary data on whether the drug adalimumab (also called Humira) can decrease pain and stiffness, improve quality of life, and is safe in people with mucopolysaccharidosis type I, II, or VI. In this study people will be randomly assigned to one of two groups. One group will be treated with adalimumab the first 16 weeks of the study and then with a saline injection for the last 16 weeks of the study. The other group will start with the saline injection for 16 weeks and then switch to adalimumab for the last 16 weeks. The study subject and the study doctor and study coordinator will not know what group a subject is in until the study is done. Adalimumab is given as an injection, just under the skin, every 2 weeks. Both groups will have blood drawn at a screening visit, and then 7 more times over the 32 week study. There will be safety labs done (liver and immune function tests). Other safety tests include a chest X-ray and screening for tuberculosis exposure - these will be done at the screening visit and later in the study if there is concern for tuberculosis exposure or a persistent cough. The following will also be done at screening, the first, middle, and last study visits: 1) a pregnancy test in all girls 8 and older, 2) questionnaires that ask about pain, how MPS impacts social and physical function, and other quality of life questions, 3) height and weight. Finally, a physical exam, that includes for children and adolescents a check of where they are in puberty, will be done by a study physician at the first, middle, and last visits. There are risks to taking adalimumab that include redness and pain where the injection is given, a decreased ability to fight off infections, and others. The safety tests are designed to identify and decrease the risk associated with adalimumab. The study physicians believe that the potential benefit of adalimumab on pain, quality of life, and other MPS related problems outweigh the potential risks of treatment.

DETAILED DESCRIPTION:
This is a randomized, pilot study consisting of a 32-week, crossover, double-blind, placebo-controlled treatment phase of subjects with Mucopolysaccharidosis (MPS) types I, II or VI treated with enzyme replacement therapy (ERT) and/or hematopoietic cell transplantation (HCT). Subjects will be treated with adalimumab (group 1) or placebo (group 2) for 16 weeks (i.e., 8 doses) then cross over to the other group for 16 weeks. Subjects will be treated with adalimumab (20 mg [weight 15-<30 kg] or 40 mg [weight ≥30 kg] administered subcutaneously [subQ] every other week) or placebo for 16 weeks, then cross-over to the other group for 16 weeks. Laboratory evaluations and Children's Health Questionnaire - Parent Form 50 (CHQ-PF50) for subjects <18 years of age or the Medical Outcomes Study Short Form-36 (SF-36) for subjects ≥18 years will be assessed at Week 16 and 32 to evaluate early treatment safety and efficacy. Safety will be assessed with laboratory evaluations at 4, 8, 20, and 24 weeks after treatment initiation, and with study visits at week 16 and 32, Physical function will be measured by the CHQ-PF50/SF-36, joint range of motion (ROM), 6-minute walk test (6MWT), and strength testing (hand-grip dynamometer) at baseline, 16, and 32 weeks. Joint inflammation will be measured by serum markers at baseline, 16, and 32 weeks. Anthropometric measurements will also be performed at Baseline and 16 and 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPS I, II or VI;
* Treatment with ERT for ≥1 year or no ERT for ≥1 year;
* Weight ≥15 kg;
* Bodily pain reported by the CHQ-PF50 or SF-36 > 1 SD below the general population mean;
* ≥ 3 joints with limitations in motion; and
* Patient or parent/legal guardian is able and willing to provide informed consent. For patients 7 to 17 years of age, assent must also be provided.

Exclusion Criteria:

* History of HCT less than 2 years prior to enrollment;
* Immune suppression therapy less than 1 year prior to enrollment;
* Active graft versus host disease;
* Current diagnosis or history of lymphoma or other malignancy;
* Current active infection;
* History of serious opportunistic infection (e.g., bacterial [Legionella and Listeria]; tuberculosis [TB]; invasive fungal infections; or viral, parasitic, and other opportunistic infections);
* Positive TB skin test, positive chest X-ray, or a recent exposure to TB
* Congestive heart failure defined by an ejection fracture <50% measured by ECHO;
* Demyelinating disorders (e.g., central nervous system [CNS] disorders including multiple sclerosis and optic neuritis and peripheral nervous system disorders including Guillain-Barre syndrome);
* Hematologic abnormalities (e.g., pancytopenia, aplastic anemia);
* Hepatitis B infection (active or chronic carrier);
* Latex sensitivity;
* Pregnancy or breastfeeding;
* Known or suspected allergy to adalimumab or related products;
* Participation in simultaneous therapeutic study that involves an investigational study drug or agent within 4 weeks of study enrollment;
* Requirement for live vaccine exposure that would be expected to occur during the time frame of the study; or
* Any other social or medical condition that the Investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or be detrimental to the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda E Polgreen, MD, MS, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pubmed/?term=28119823

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab First, Then Placebo: Participants first received Adalimumab 20 mg subQ every other week (weight 15 to <30 kg) or 40 mg subQ every other week (weight ≥30 kg) for 16 weeks. Participants then received Placebo saline subQ (volume matching Adalimumab 20 mg or 40 mg subQ) every other week.
- Placebo First, Then Adalimumab: Participants first received Placebo saline subQ (volume matching Adalimumab 20 mg or 40 mg subQ) every other week. Participants then received Adalimumab 20 mg subQ every other week (weight 15 to <30 kg) or 40 mg subQ every other week (weight ≥30 kg) for 16 weeks.
Period: Overall Study
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15 [15 to 15] | 6 [6 to 6] | 10.5 [6 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Children's Health Questionnaire - Parent Form 50 Bodily Pain Standardized Score
Description: Children's Health Questionnaire - Parent Form 50 bodily pain (BP) standardized score for participants < 18 years of age. Range is from 0 to 100 (no units) and standardization if determined by comparison to healthy age matched children. Lower values mean increased pain. The difference of change in BP standardized score from day 0 to week 16 during adalimumab treatment minus change in BP standardized score from day 0 to week 16 during placebo treatment is reported.
Time Frame: day 0 to week 16 of treatment with adalimumab versus placebo
Population: This was a cross-over study so within-individual changes are reported.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab
Number analyzed (Participants) | 1 | 1
units on a scale | 1.4 [1.4 to 1.4] | 1.0 [1.0 to 1.0]

2. Secondary Outcome: Children's Health Questionnaire - Parent Form 50 Physical Function (PF) Standardized Score
Description: Children's Health Questionnaire - Parent Form 50 physical function (PF) standardized score for participants < 18 years of age. Range is from 0 to 100 (no units) and standardization if determined by comparison to healthy age matched children. Lower values mean decreased physical function. The difference of change in PF standardized score from day 0 to week 16 during adalimumab treatment minus change in PF standardized score from day 0 to week 16 during placebo treatment is reported.
Time Frame: Day 0 to week 16 of treatment with adalimumab versus placebo
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab
Number analyzed (Participants) | 1 | 1
units on a scale | 0 [0 to 0] | 0.4 [0.4 to 0.4]

3. Secondary Outcome: Pain Measured by the Visual Analog Scale (VAS) in the Pediatric Pain Questionnaire (PPQ)
Description: Percent of participants with a >10 mm improvement in either "how you feel now" or "worst pain you had this week" on the VA in the PPQ during adalimumab versus during placebo by either parental or subject report. Range is 0-100 mm; lower number means less pain.
Time Frame: Day 0 to week 16 of treatment with adalimumab versus placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

4. Secondary Outcome: Range of Motion - Bilateral Shoulder, Elbow, Hip, Knee
Description: Number of joints with a >5 degree more positive change during 16 weeks of adalimumab versus 16 weeks of placebo. A total of eight joints were measured.
Time Frame: Day 0 to week 16 of treatment with adalimumab versus placebo
Measure: Number; unit: joints
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab
Number analyzed (Participants) | 1 | 1
joints | 7 | 5

5. Secondary Outcome: Anti-ERT Antibodies
Description: Anti-laronidase antibodies for subjects with MPS I. Anti-idursulfase antibodies for subjects with MPS II.
Time Frame: Day 0 to week 16 of treatment with adalimumab versus placebo
Population: No participants had anti-ERT antibodies
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab First, Then Placebo | Placebo First, Then Adalimumab
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Adalimumab: 20 mg subQ every other week (weight 15 to <30 kg) 40 mg subQ every other week (weight ≥30 kg).
  Adalimumab: Subjects will be treated with adalimumab (20 mg [weight 15-<30 kg] or 40 mg [weight ≥30 kg] administered subcutaneously [subQ] every other week) or placebo for 16 weeks, then cross-over to the other group for 16 weeks.
- Placebo: Saline placebo injection
  Placebo: Saline placebo
Arm/Group | Adalimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=2) | Placebo (N=2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Resolved after 2 days without intervention
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Resolved by 2 week recheck without intervention
Mood lability (Psychiatric disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Injection site erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small pilot study of 2 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No